CLINICAL TRIAL: NCT06897436
Title: "EUmetriosis: Transforming Endometriosis Care in Europe: an Integrated Approach to Enhance Understanding, Diagnosis, Tailored Management and Patient Empowerment
Brief Title: Characterization of Immune Cells and Their Secreted Cytokines in Endometriosis Patients
Acronym: EUmetriosis
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Lublin (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Iwona Wertel, professor, Medical University of Lublin
Other Study IDs: 101157146; Project 101157146-EUmetriosis (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: endometriosis; dermoid cyst; immune system
MeSH Terms: conditions — Endometriosis; Dermoid Cyst

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — peripheral blood, menstrual effluent/blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: pre-menopausal adult women with clinically and/or ultrasound-diagnosed endometriosis, age between 18 and 40 years, with regular menstruation, without autoimmune diseases, without malignant diseases

SUMMARY:
The EUmetriosis project aims to address the most important unmet needs of endometriosis sufferers to advance patient care. The objectives cover all main aspects of disease management, including elucidating the pathogenesis, diagnosing the condition promptly and efficiently, facilitating care by implementing self-management strategies, raising awareness and promoting policy changes. The objectives comprise individual yet intersecting pieces of a puzzle which, when positioned correctly, can immensely improve disease perception and understanding to enhance patient care. The project will prioritise the needs and wants of modern-day patients, focused on providing easily accessible and noninvasive therapeutic options. Combining all these elements in a well-coordinated project is pivotal to relieving the heavy burden endometriosis places on European society as a whole.

DETAILED DESCRIPTION:
EUmetriosis will generate new knowledge in the field of endometriosis, its drivers and consequences, as well as biological determinants, which will result in a better understanding of endometriosis pathogenesis and the factors involved. Specifically, the project will assess the role of the immune cells, diet, cognitive behaviour and other related factors in disease pathogenesis, and develop strategies on how to alleviate endometriosis-associated pain, enhance quality of life and improve outcomes for patients. The knowledge base (like the association between nutrition, epigenetics, the microbiome and endometriosis) and methodologies generated within the project will drive the fields of gynaecology, primary care, pain medicine, urology and gastroenterology forward. Finally, through the collection of evidence for effective self-management strategies, the project will pave the path for more patient-tailored health policies. The project aims to link different stakeholder groups involved in this field, like clinicians, patients, healthcare insurers/payers and other researchers in women's health. With this multidisciplinary consortium, EUmetriosis will maximise its impact by creating therapeutic and diagnostic endometriosis solutions best suited to real-world applications, with a clear strategy for implementation.

ELIGIBILITY:
Inclusion Criteria:

* Women with a clinical and/or ultrasound diagnosis of endometriosis who are candidates for surgery
* Age between 18 and 50 years
* Pre-menopausal status
* Experiencing regular menstruation
* Willing to collect menstrual effluent
* Signature of informed consent to the study

Exclusion Criteria:

* Age below 18 years
* Post-Menopausal status
* Presence of Crohn's disease
* Presence of Ulcerative Colitis
* Presence of short bowel syndrome or another chronic inflammatory disease
* Use immunosuppressive medication
* Receiving contraceptive hormone therapy
* Pregnant
* Presence/history of malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The University Clinical Hospital No.4 and No.1, 1 Military Clinical Hospital in Lublin SPZOZ
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Alterations in immune system cell phenotype and activity associated with endometriosis. | The collection of peripheral blood samples will be done at a single time point before the surgery. Collection of menstrual effluent in the form of a menstrual cup on the 2nd day of the menstrual cycle.
  High-dimensional flow cytometry (FACS) will be done to analyse immune cells such as Myeloid derived suppressor cells (MDSC) along with the expression of co-inhibitory molecules on their surface. Functional parameters crucial to MDSCs activity will be than investigated (ARG1, IDO, NOS2, IL-10, TGFβ) in endometriosis patients and in the control group, to evaluate their immune profile. Also Natural Killer (NK) cells and γδ T cells along with co-inhibitory (TIGIT, LAG-3, TIM-3,PD-1) and co-stimulatory (CD16, NKG2D and OX40, CD226 (DNAM-1) immune checkpoints expression will be characterised, to determine any differences between patients with and without endometriosis. Functional parameters crucial to NK cells and γδ T lymphocytes activity will be also investigated (CD3ζ (CD247), granzyme B, perforin, and IFN-γ).
Alterations in the level of inflammatory and immunosuppressive cytokines associated with endometriosis. | The collection of peripheral blood samples will be done at a single time point before the surgery. Collection of menstrual effluent in the form of a menstrual cup on the 2nd day of the menstrual cycle.
  High-dimensional flow cytometry and ELISA will be done to analyse the level of the soluble forms of immune checkpoint (sTIM-3, sGal-9, sTIGIT, sCD155, LAG-3, sOX40L, sOX40) and soluble factors (IL-1beta, IL-6, IL-8, IL-12p70, IL-2, IL-4, IL-6, IL-10, IL-17A, TNF-α, and IFN-γ) in plasma of patients with endometriosis and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jarogniew Łuszczki, professor, Study Director — UNIWERSYTET MEDYCZNY W LUBLINIE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CORDIS belongs to the Research and Innovation community platform of the European Commission and complements the Funding and tender opportunities website, where there is possibility to apply for funding and search for partners. — https://cordis.europa.eu/project/id/101157146